CLINICAL TRIAL: NCT01859195
Title: Monoclonal Antibody-based Multipurpose Microbicides
Acronym: Project WIND
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: Boston University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIDS-ES-ID-11941; U19AI096398 (NIH)
Record Dates: First submitted 2013-05-14; First posted 2013-05-21 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: HIV; Sexually Transmitted Infections (STI)
Keywords: HIV/STI; Prevention; Microbicides, Topical
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Focus Group Stage: ~20-24 participants, to comprise 3-6 focus groups
- Cognitive Interview Stage: ~12-16 participants in individual cognitive interviews

SUMMARY:
The purpose of this project is to explore women's thoughts, opinions, and ideas about vaginal products. The investigators will ask women to help design the best strategy for applying a vaginal product using a specific kind of applicator. The investigators want to identify designs that women think would be easy to prepare and insert. Women's thoughts and opinions will help researchers develop new products called microbicides that may protect against HIV and other sexually transmitted diseases, that are easy to use, and that will be acceptable to women who use them. If researchers can make products that are easy to use and that women like to use, the products will be used more often, and more infections will be prevented.

Women who enroll in the project will either participate in a focus group with approximately 3-7 other women or a one-on-one cognitive interview. All participants will complete a brief questionnaire. Some women may enroll in both stages.

Each focus group will take approximately 1.5-2.5 hours. Group leaders will talk to women about their experiences using vaginal products and will provide participants with study products to look at and touch. All participants will be asked to come up with ideas of how to make the products easy to use and acceptable to women who use them. Group leaders will encourage discussion about the different designs. After this, group leaders will talk about a specific type of microbicide and ask women about their opinions. In particular, researchers and participants will talk about the language that would be best understood by women who would use these products or be in studies to evaluate them.

Each cognitive interview will take approximately 1.5-2.5 hours. Each participant will be asked about different product designs and application instructions, and will be asked her thoughts, opinions, and potential concerns about each. She will also evaluate sample language that will be used to help women understand the products and how to use them.

ELIGIBILITY:
Inclusion Criteria:

Women who:

* are between the ages of 18 and 45 at prescreening
* report vaginal sex with a man in the past 12 months at prescreening
* report negative pregnancy status and no intention to become pregnant during the course of the study
* report negative or unknown HIV status, and
* are willing and able to provide informed consent.

Exclusion Criteria:

Women who:

* self-report being pregnant, or intention to become pregnant during the course of the study
* self-report being HIV-positive
* self-report an allergy or sensitivity to vaginal contraceptive film (VCF), nonoxynol-9 (N9), or product(s) containing N9
* are unable or unwilling to give informed consent, or
* have any condition that, in the opinion of the project leader or principle investigator, would compromise the participant's ability to participate in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females who are 18-45 years old, HIV negative or unknown (self report), non-pregnant and not intending to get pregnant (self report), and report vaginal sex with a man in the past 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2022-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Morrow, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital - ReproHelath Team, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited May-Aug 2013 (RI, MA USA) via call-lists, flyers, ads, internet/social media, clinics, CBOs, word-of-mouth. Volunteers complete prescreen survey. If eligible, each invited to participate in either (1) focus group or (2) individual cognitive interview (first ~20-24 for focus groups; remaining ~12-16 for interviews after FGs began).
Period: Overall Study
Arm/Group | Focus Group Stage | Cognitive Interview Stage
Started | 24 | 12
Completed | 24 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Focus Groups: Focus Groups
- Cognitive Interviews: Cognitive Interviews
- Total: Total of all reporting groups
Arm/Group | Focus Groups | Cognitive Interviews | Total
Number analyzed (Participants) | 24 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 12 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 12 | 36
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 23 | 8 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 15 | 8 | 23
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants: Comprehension of Study Product
Description: Focus groups captured participant understandings (in narrative form) of plant-produced monoclonal antibodies, how they come about, how they are manufactured, how they differ from other anti-HIV actives, etc. Participant-derived language informed development of study materials, including study product instruction sheets and informed consent materials and documents.
  Cognitive Interview assessed Participant comprehension of language used in insertion instruction materials, and monoclonal antibody education and informed consent materials.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants: Focus Group: Number of participants in focus group stage
- Number of Participants: Cognitive Interviews: Number of participants in cognitive interview stage
Arm/Group | Number of Participants: Focus Group | Number of Participants: Cognitive Interviews
Number analyzed (Participants) | 24 | 12
Participants | 24 | 12

2. Other Pre Specified Outcome: Number of Participants: Drug Delivery Systems Evaluations
Description: Members of focus groups evaluated various drug delivery system designs, to determine final design to move forward with in development
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants: Focus Groups: number of participants who completed focus group stage
- Number of Participants: Cognitive Interviews: number of participants who completed cognitive interview stage
Arm/Group | Number of Participants: Focus Groups | Number of Participants: Cognitive Interviews
Number analyzed (Participants) | 24 | 12
Participants | 24 | 12

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Focus Groups | Cognitive Interviews
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 0/24 | 0/12

LIMITATIONS AND CAVEATS:
This is a formative qualitative data study, designed to gather narrative participant-relevant information related to study product development and evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No